CLINICAL TRIAL: NCT00929656
Title: Combining Neural and Behavioral Therapies to Enhance Stroke Recovery
Brief Title: Combined Neural and Behavioral Therapies to Enhance Stroke Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B6862-W
Record Dates: First submitted 2009-06-25; First posted 2009-06-29 (Estimated); Results first posted 2017-07-05 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Stroke
Keywords: Rehabilitation; Neurophysiology; Upper Extremity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real rTMS (Experimental): Real rTMS + unimanual paretic UE training
  Interventions: Procedure: Real rTMS; Procedure: Unimanual paretic UE Training
- Sham rTMS (Active Comparator): Sham rTMS + unimanual paretic UE training
  Interventions: Procedure: Sham rTMS; Procedure: Unimanual paretic UE Training

INTERVENTIONS:
Procedure: Real rTMS — rTMS application to lesioned hemisphere; 10 Hz, 1000 pulses
  Arms: Real rTMS
Procedure: Sham rTMS — sham rTMS application to lesioned hemisphere; 10 Hz, 1000 pulses
  Arms: Sham rTMS
Procedure: Unimanual paretic UE Training — UE exercise for 4 hours (two hours 1:1 with therapist and two hours independent at home) for 16 sessions (4 sessions/week for 4 weeks)

SUMMARY:
Stroke is the leading cause of long-term disability in this country with more than 1 million Americans reporting difficulty with daily activities. Loss of independence in self-care tasks is primarily due to limited recovery of the arm. This study will determine if the addition of Transcranial Magnetic Stimulation (TMS) to excite the lesioned hemisphere (side of the brain affected by the stroke), to progressive functional task exercise either of the weakened arm alone or of both arms together will improve arm recovery to a greater degree than one of these two types of arm exercise alone. Individuals post-stroke will participate in 16 sessions of 1) arm rehabilitation alone (with the weaker arm only or with both arms together) or 2) arm rehabilitation plus TMS. The investigators will assess arm movement ability and function immediately following the 4-week intervention and at a 30-day follow-up to determine retention of immediate gains. The investigators hypothesize that those who receive TMS as an adjuvant will have improved arm movement ability than those who only exercise.

DETAILED DESCRIPTION:
Limited recovery of upper extremity (UE) function post-stroke continues to be one of the greatest challenges faced in neurorehabilitation. There is an urgent unmet need to identify effective approaches to drive UE recovery in this population. In response to this challenge, the overall purpose of this proposed research plan is to develop rehabilitation interventions that restore UE motor recovery. Contemporary approaches to motor rehabilitation are based on evidence that behavioral experience drives cortical reorganization following neural injury. Although the rationale of driving the damaged motor cortex by focused training of the paretic UE appears straightforward, and has historically been the focus of rehabilitation, functional recovery remains limited. There remains a gap between this central neurobiological change and a meaningful behavioral change. There is a need, therefore, to augment or potentiate behavioral experience. This proposal will address this gap by examining two potential drivers of the lesioned hemisphere: 1) the non-lesioned hemisphere via engagement of the unaffected UE in behavioral training and 2) stimulation of the lesioned hemisphere via repetitive Transcranial Magnetic Stimulation (rTMS). This proposal builds on the foundation of the applicant's previous work which suggested that the contralesional, intact, hemisphere could be used to drive the lesioned hemisphere through bimanual movement. Additionally, it is possible to drive the lesioned hemisphere externally using rTMS to enhance cortical stimulation. Thus, pairing externally-driven enhancement of cortical excitability with internally-driven activation of the intact hemisphere during bilateral movements could combine to further increase excitability in the lesioned hemisphere and manifest improved movement capability of the paretic UE. The fundamental hypothesis guiding this proposal is that increased excitability of the lesioned cortex will improve behavioral function of the paretic UE post-stroke. To investigate the overall hypothesis the investigators will examine these drivers of cortical excitability and their role in UE recovery by addressing the following aims:

Specific Aim 1. Determine the magnitude of difference in central and behavioral changes in individuals with post-stroke hemiparesis randomized to a bilateral versus unilateral UE motor training program.

Specific Aim 2a. Determine the magnitude of difference in central and behavioral changes in individuals with post-stroke hemiparesis randomized to behavioral UE training compared to behavioral UE training + rTMS.

Specific Aim 2b. Determine the differential effects of rTMS on bilateral behavioral training compared to unilateral behavioral training as measured both centrally and behaviorally in individuals with post-stroke hemiparesis Post-stroke upper limb paresis and resultant loss of functional ability continues to present a barrier to those post-stroke in returning to full societal participation. Interventions that directly target the mechanism of hemiparesis, including decreased excitability of the lesioned hemisphere, are most likely to promote true recovery as opposed to the oft observed functional compensation in these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1st stroke > 6 months
* Sub-cortical stroke confirmed with CT or MRI
* Passive range of motion in bilateral shoulder and elbow within functional limits
* UE Fugl-Meyer shoulder/elbow subcomponent score between 15 - 25
* 18-80 years of age

Exclusion Criteria:

* Use of medications that may lower seizure threshold
* History of epilepsy, brain tumor, learning disorder, mental retardation, drug or alcohol abuse, dementia, major head trauma, or major psychiatric illness
* evidence of epileptiform activity on EEG obtained before beginning treatment
* history or radiographic evidence of arteriovenous malformation, intracortical hemorrhage, subarachnoid hemorrhage, or bilateral cerebrovascular disease,
* history of cortical stroke
* history of implanted pacemaker or medication pump, metal plate in skull, or metal objects in the eye or skull
* pregnancy
* pain in either upper extremity that would interfere with movement
* unable to understand 3-step directions
* orthopedic condition in back or UE or impaired corrected vision that would alter kinematics of reaching

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-02-01; Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorian Kay Rose, PhD MS BS, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Malcom Randall VA Brain Rehabilitation Research Center database from 2/1/13-9/30/15
Groups:
- Unimanual UE Training + Real rTMS: Unimanual Upper Extremity (UE) training + repetitive Transcranial Magnetic Stimulation (rTMS)
  Unimanual UE training + rTMS: rTMS application to lesioned hemisphere followed by unimanual (paretic) UE functional task practice (2 hours) for 16 sessions (4 sessions/week for 4 weeks)
- Unimanual UE Training + Sham rTMS: Unimanual Upper Extremity (UE) training + sham repetitive Transcranial Magnetic Stimulation (rTMS)
  Unimanual UE training + sham rTMS: sham rTMS application to lesioned hemisphere followed by unimanual (paretic) UE functional task practice (2 hours) for 16 sessions (4 sessions/week for 4 weeks)
Period: Overall Study
Arm/Group | Unimanual UE Training + Real rTMS | Unimanual UE Training + Sham rTMS
Started | 13 | 9
Completed | 13 | 8
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Unimanual UE Training + Real rTMS: Participants randomized to the Experimental Arm received real rTMS (1000 pulses) to their ipsilesional hemisphere followed by two hours of paretic arm functional task practice administered/supervised by a physical therapist.
- Unimanual UE Training + Sham rTMS: Participants randomized to the Placebo Arm received sham rTMS to their ipsilesional hemisphere followed by two hours of paretic arm functional task practice administered/supervised by a physical therapist.
- Total: Total of all reporting groups
Arm/Group | Unimanual UE Training + Real rTMS | Unimanual UE Training + Sham rTMS | Total
Number analyzed (Participants) | 13 | 9 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (10.0) | 59.4 (8.2) | 60.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 12 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 11 | 5 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 9 | 22
Time Post-Stroke [Mean (Standard Deviation); unit: months] — The amount of time, in months, between stroke onset and entrance into the study.
  months | 44.0 (95.6) | 33.3 (25.9) | 39.6 (74.2)

OUTCOME MEASURES:

1. Primary Outcome: Wolf Motor Function Test Change
Description: Change, in seconds, between Pre-intervention and post-intervention (4 wks following pre-intervention). The time to complete 15 separate upper extremity functional tasks are recorded. These 15 separate timed events are averaged to provide one time, in seconds. This is considered an Activity Measure on the WHO ICF model.
Time Frame: Change between Pre-intervention (baseline) to Post-intervention (4 wks following pre-intervention)
Measure: Mean (Standard Error); unit: seconds
Groups:
- Unimanual UE Training + Real rTMS: Unimanual UE training + rTMS
  Unimanual UE training + rTMS: rTMS application to lesioned hemisphere followed by unimanual (paretic) UE functional task practice (2 hours) for 16 sessions (4 sessions/week for 4 weeks)
- Unimanual UE Training + Sham rTMS: Unimanual UE training + sham rTMS
  Unimanual UE training + sham rTMS: sham rTMS application to lesioned hemisphere followed by unimanual (paretic) UE functional task practice (2 hours) for 16 sessions (4 sessions/week for 4 weeks)
Arm/Group | Unimanual UE Training + Real rTMS | Unimanual UE Training + Sham rTMS
Number analyzed (Participants) | 13 | 9
seconds | 1.6 (1.1) | 1.8 (1.2)

2. Secondary Outcome: Upper Extremity Fugl-Meyer Motor Assessment Change
Description: Change in Score from Pre-intervention to Post-Intervention. This outcome measures arm motor control; the ability to move outside of pathologic synergistic patterns. It is a measure of impairment in Body Structure/Function. Total score ranges from 0-66, with 0 indicative of no movement and 66 considered normal motor control.
Time Frame: Change Between Pre-intervention (baseline) to Post-intervention (4 wks following pre-intervention)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Unimanual UE Training + Real rTMS | Unimanual UE Training + Sham rTMS
Number analyzed (Participants) | 13 | 9
units on a scale | 5.8 (1.4) | 5.8 (1.1)

3. Secondary Outcome: Grip Strength Change
Description: Change in Paretic hand grip strength from pre- to post-intervention. Grip strength measured by hand-held dynamometer. An average of 3 5-second trials was used for analysis.
Time Frame: Change between Pre-intervention (baseline) to Post-intervention (4 wks following pre-intervention)
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Unimanual UE Training + Real rTMS | Unimanual UE Training + Sham rTMS
Number analyzed (Participants) | 13 | 9
kilograms | 1.1 (2.0) | 1.3 (2.4)

4. Secondary Outcome: Motor Activity Log - Amount of Use Change
Description: Self-Report Amount of Use of Paretic UE to complete 30 functional tasks. Each task is reported on a 0-5 scale with "0" representing "did not use my paretic hand at all for that task" and "5" representing "I used my paretic hand as much as before the stroke to complete that task." A "5" on each task would be considered "normal."
Time Frame: Change Between Pre-intervention (baseline) to Post-intervention (4 wks following pre-intervention)
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Unimanual UE Training + Real rTMS | Unimanual UE Training + Sham rTMS
Number analyzed (Participants) | 13 | 9
Units on a scale | 1.3 (0.3) | 1.2 (0.3)

5. Secondary Outcome: Motor Activity Log - How Well Change
Description: Self-Report of How Well paretic UE performed completing 30 functional tasks. Each task is reported on a 0-5 scale with "0" representing "Unable to use my paretic hand to perform that task" and "5" representing "My paretic hand performs that task as well as it did before the stroke." A "5" on each task would be considered "normal."
Time Frame: Change between Pre-intervention (baseline) to Post-intervention (4 wks following pre-intervention)
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Unimanual UE Training + Real rTMS | Unimanual UE Training + Sham rTMS
Number analyzed (Participants) | 13 | 9
Units on a scale | 1.1 (0.3) | 1.2 (0.4)

ADVERSE EVENTS:
Groups:
- Unimanual UE Training + Real rTMS: Unimanual UE training + rTMS
  Unimanual UE training + rTMS: rTMS application to lesioned hemisphere followed by unimanual (paretic) UE exercise (100 repetitions) for 16 sessions (4 sessions/week for 4 weeks)
- Unimanual UE Training + Sham rTMS: Unimanual UE training + sham rTMS
  Unimanual UE training + sham rTMS: sham rTMS application to lesioned hemisphere followed by unimanual (paretic) UE exercise (100 repetitions) for 16 sessions (4 sessions/week for 4 weeks)
Arm/Group | Unimanual UE Training + Real rTMS | Unimanual UE Training + Sham rTMS
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/9
Other Adverse Events (participants affected / at risk) | 0/13 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes